CLINICAL TRIAL: NCT06284707
Title: Effect of an Adapted Rhythmic Gymnastics Training Program in Children With Down Syndrome
Brief Title: Effect of Rhythmic Gymnastics Training in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: Rhythmic_PAU_2024
Record Dates: First submitted 2024-02-02; First posted 2024-02-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-02

CONDITIONS: Physical Conditioning, Human
Keywords: rhythmic gymnastics; disability; gymnastics training; down syndrome; child
MeSH Terms: conditions — Motor Activity; Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The care provider will be responsible for administering the training program. Two different people will develop swimming training and rhythmic gymnastics training. Each participant will be assigned a code. The researcher will process the data with the code of each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- swimming training (Other): Participants complete 2 swimming training sessions per week. Total program time 10 weeks
  Interventions: Other: swimming training
- swimming training and rhythmic gymnastics training (Experimental): Participants perform 2 swimming training sessions per week and 2 rhythmic gymnastics training sessions.
  Total program time 10 weeks
  Interventions: Other: swimming training; Other: rhythmic gymnastics training

INTERVENTIONS:
Other: swimming training — 2 sessions per week of swimming training
Other: rhythmic gymnastics training — 2 training sessions of rhythmic gymnastics
  Arms: swimming training and rhythmic gymnastics training

SUMMARY:
Some of the clinical characteristics of people with Down syndrome (DS) are orthopedic, cardiovascular, neuromuscular, visual, cognitive and perceptual disorders, which directly affect the quality of their movements. Children with DS often have a sedentary lifestyle or low levels of physical activity which exacerbates problems related to obesity and overall physical health. Therefore, the practice of physical exercise in this type of population is essential to improve their health-related physical fitness. The aim of this study was to analyze the influence of an adapted rhythmic gymnastics training program on body composition, tendon architecture and stiffness, and physical capacity in children with DS.

DETAILED DESCRIPTION:
Children with DS with medium to moderate intellectual disabilities are required to participate. Participants will complete 10 weeks of training, two days per week. They will be divided into two groups: the Control Group will receive two swimming sessions per week and the Experimental Group will receive two swimming sessions plus two rhythmic gymnastics sessions. Before and after the application of the program, the following will be evaluated: body composition by Inbody 720, muscular architecture and elastography by Logiq® S8 ultrasound scanner and tendon stiffness by Myoton® Pro portable myotonometer. The tendons to be studied will be the Achilles tendon and the patellar tendon.

ELIGIBILITY:
Inclusion Criteria:

* Disabiluty: mild to moderate

Exclusion Criteria:

* Any contraindication to exercise
* Severe or profound intellectual disability
* Musculoskeletal disorders that prevented completion of the tests

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Body composition | "baseline" and "immediately post intervention"
  Body compisition will be assessed with the Inbody 720 (Bioespace, Seoul, Korea). In this test body mass (BM; kg), muscle mass (MM; kg), fat mass (FM; kg), lean mass (LM; kg), fat-free mass (FF; kg)
Tendon thickness | "baseline" and "immediately post intervention"
  Tendon thickness will be evaluated with the Logiq® S8 ultrasound machine (GE Healthcare, Milwaukee, WI).
Stiffness tendon | "baseline" and "immediately post intervention"
  Stiffness tendon will be evaluated with Myoton® Pro hand-held myotonometer (Myoton AS, Tallinn, Estonia). In this test, the mechanical properties of the Achilles tendon will be measured.
Hamstrings flexibility | "baseline" and "immediately post intervention"
  Hamstrings flexibility will be evaluated with Seat and Reach Test (Fabrication Enterprises Inc., USA).
body mass index | "baseline" and "immediately post intervention"
  Body mass index (BMI; kg/m2) will be calcultated from body mass and height
visceral fat area | "baseline" and "immediately post intervention"
  visceral fat area (area; cm2) will be assessed with the Inbody 720 (Bioespace, Seoul, Korea).
metabolism | "baseline" and "immediately post intervention"
  metabolism (MET; kcal) will be assessed with the Inbody 720 (Bioespace, Seoul, Korea).
tendon elastography | "baseline" and "immediately post intervention"
  Tendon elastography will be evaluated with the Logiq® S8 ultrasound machine (GE Healthcare, Milwaukee, WI).
balance | "baseline and "immediately post intervention"
  Balance will be evaluated with the Biodex Balance System stability system (Biodex Medical Systems Inc., USA).
functional capacity | "baseline" and "immediately post intervention"
  Functional capacity of the lower body wll be evaluated with Sit to Stand Test adapted.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Abián-Vicén, PhD, Study Director — University of Castilla-La Mancha
Locations (1):
- Universidad de Castilla La Mancha, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No